CLINICAL TRIAL: NCT05477264
Title: Phase II Study of Concurrent Tislelizumab and Radiotherapy for Treatment-naïve, Newly Diagnosed Low-risk Extranodal NK/T-cell Lymphoma, Nasal Type
Brief Title: Concurrent Tislelizumab and Radiotherapy in Newly Diagnosed Extranodal NK/T-cell Lymphoma, Nasal Type
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Won Seog Kim (Other)
Responsible Party: Sponsor-Investigator, Won Seog Kim, Clinical Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-03-082
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab therapy (Experimental): Induction therapy: Tislelizumab combined with radiation
  Maintenance therapy(after termination of combination therapy)
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Induction therapy: Tislelizumab combined with radiation
  * Tislelizumab: 200mg, IV at 3-week intervals combined with radiotherapy.
  * Radiotherapy: 400Gy/20 fractions
  Maintenance therapy(after termination of combination therapy)
  * Tislelizumab: 200mg IV at 3-week intervals for up to 2 years until disease progression or intolerance.

SUMMARY:
This clinical trial intends to analyze the efficacy of PD-1 inhibitor combined with radiotherapy for newly diagnosed NK/T-cell lymphoma. The investigational product in this clinical trial is tislelizumab, a PD-1 inhibitor.

As a rationale for using PD-1 inhibitors in patients with NK/T-cell lymphoma, their efficacy has been proved several times mostly in patients with relapsed NK/T-cell lymphoma.

Patients with low-stage NK/T-cell lymphoma usually receive high-concentration cytotoxic chemotherapy combined with radiotherapy, with treatment response rates of approximately 60 to 80%, but 80-90% of them experience hematological and non-hematologic toxicities during treatment.

Therefore, this study intends to determine the efficacy and safety of PD-1 inhibitor(Tislelizumab) combined with radiotherapy as a first-line therapy compared with pre-existing cytotoxic chemotherapy combined with radiotherapy in patients with NK/T-cell lymphoma with low stage and International Prognostic Index.

DETAILED DESCRIPTION:
This clinical trial intends to analyze the efficacy of PD-1 inhibitor combined with radiotherapy for newly diagnosed NK/T-cell lymphoma. The investigational product in this clinical trial is tislelizumab, a PD-1 inhibitor.

As a rationale for using PD-1 inhibitors in patients with NK/T-cell lymphoma, their efficacy has been proved several times mostly in patients with relapsed NK/T-cell lymphoma.

However, a tumor-immune microenvironment(TIME) analysis at our institution confirmed that patients with relapsed or refractory NK/T-cell lymphoma had a peritumoral microenvironment with suppressed activity of T cells and macrophages (immune suppression, IS), in which case the efficacy of PD-1 inhibitor decreased compared to a more immune-active microenvironment (immune evasion or immune tolerance, IE or IT). On the other hand, most patients who were newly diagnosed with NK/T-cell lymphoma had a peritumoral microenvironment with active T cells and macrophages(IE or IT).

Patients with low-stage(Stage IE or IIE) NK/T-cell lymphoma usually receive high-concentration cytotoxic chemotherapy combined with radiotherapy, with treatment response rates of approximately 60 to 80%, but 80-90% of them experience grade 3 or 4 hematological and non-hematologic toxicities during treatment.

Therefore, based on the tumor microenvironment of NK/T-cell lymphoma, this study intends to determine the efficacy and safety of PD-1 inhibitor(Tislelizumab) combined with radiotherapy as a first-line therapy compared with pre-existing cytotoxic chemotherapy combined with radiotherapy in patients with NK/T-cell lymphoma with low stage and International Prognostic Index.

ELIGIBILITY:
Inclusion Criteria:

1. Histologicallly diagnosed extranodal NK/T-cell lymphoma
2. No history of prior treatment
3. Stage IE/IIE(cases involving the nasal cavity, nasopharynx, and oral cavity only)
4. International prognostic index(PINK, PINK-E risk score): 0-1
5. 19 years and older
6. ECOG PS: 0-2
7. AT least one measurable and assessable lesion at least 1.5cm in size on CT or PET/CT scan
8. Adequate bone marrow function, as defined by the following laboratory values(If cytopenia is associated with bone marrow involvement, the subject is excluded):

   * Absolute neutrophil > 1,500/mm3
   * Hemoglobin > 9.0g/dL
   * Platelet > 75,000/mm3
9. Adequate organ function, as defined by the following laboratory values

   * Total bilirubin, AST/ALT < 3xULN
   * Serum creatinine ≤ 2.0mg/dL
10. Voluntary written informed consent to undergo chemotherapy and radiotherapy
11. Female subjects are required to meet the following criteria:

    * Pregnancy test: For women of childbearing potential, a negative serum or urine pregnancy test at screening
    * Contraception: For both male and female subjects, use of highly effective contraception throughout the study period and, if at risk of pregnancy, for at least 6 months after the last dose of the study treatment
12. Having tumor tissue sample in storage available for targeted sequencing

Exclusion Criteria:

1. History of prior treatment(chemotherapy, radiotherapy, or targeted therapy) to treat extranodal NK/T-cell lymphoma
2. Stage III/IV at diagnosis or stage IE-IIE with extranodal(cutaneous, soft tissue, gastrointestinal, brain, spinal cord, bone marrow, etc.)
3. International prognostic index(PINK, PINK-E): ≥ 2
4. Has a concomitant malignancy or had a malignancy(except for appropriately treated basal or squamous cell carcinoma or cervical carcinoma in situ) in the last 3 years prior to initiation of the study treatment
5. Underwent a major surgery within 21 days prior to initiating the study treatment, or has not recovered from serious side effects of surgery
6. Concomitant use of immunosuppressants, except for the following:

   * Intranasal, inhaled, or topical steroid, or local steroid injection(such as intra-articular injection)
   * Physiological dose ≤ 10mg/day of prednisone or equivalent doses of systemic corticosteroid
   * Premedication with steroids to prevent hypersensitivity reaction(such as premedication prior to a CT scan). At the discretion of the investigator, the use of prednisolone at ≥ 10mg for adrenal insufficiency may be acceptable
7. Clinically significant, or active, cardiovascular disease

   * Cerebrovascular accient/stroke: within 6 months prior to study entry
   * Myocardial infarction: within 6 months prior to study entry
   * Unstable angina, congestive heart failure(New York Heart Association class ≥II), or serious cardiac arrhythmias requiring medication, including any of the following

     * Left ventricular ejection fraction(LVEF) < 50% as measured by echocardiography
     * QTc>480msec(using the QTcF formula) on ECG at screening
     * unstable angina
     * ventricular arrhythmias except for benign premature ventricular contraction
     * medically uncontrolled supraventricular and nodal arrhythmias
     * conduction abnormality requiring a pacemaker
     * valve disease with documented cardiac dysfunction
8. Other concomitant severe and/or uncontrolled medical conditions(e.g., uncontrolled diabetes mellitus, chronic pancreatitis, active chronic hepatitis, etc.) that the investigator considers would preclude the subjects's participation in the clinical trial. Other severe acute or chronic medical conditions include colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis, or psychiatric conditions, including recent(in the last 1 year) or active suicidal thoughts or behaviors: or laboratory abnormalities the, in the investigator's opinion, may increase the risk associated with participation in the clinical trial or study treatment, or that may interfere with the interpretation of clinical trial results.
9. Active infection requiring ststemic therapy
10. Active autoimmune disease that may be exacerbated upon administration of immunostimulants. However, subjects with type I diabetes mellitus, vitiligo, psoriasis, or hypothyroidism or hyperthyroidism not requiring immunosuppressive treatment are eligible
11. Incapable of understanding or complying with clinical trial instructions and requirements, or have a history of noncompliance with medical therapy
12. Pregnant or nursing(breastfeeding) women. Pregnancy is defined as the condition of a woman form pregnancy as confirmed by positive serum hCG laboratory test(>5mIU/mL) to termination of pregnancy.
13. Live vaccination is prohibited, except for influenza and COVID vaccines are allowed, within 2 weeks prior to the first dose of tislelizumab and during clinical trial participation, and inactivated vaccines are allowed.
14. Hepatitis B virus(HBV) related liver disease, such as the following:

    * Chronic hepatitis with cirrhosis
    * HBV reactivation(However, hepatitis B surface antigen positive subjects who are asymptomatic and do not require treatment can be enrolled at the discretion of the investigator)
    * Hepatitis B virus(HBV) infection at screening(HBV surface antigen-positive and HBV DNA positive)
    * Hepatitis C virus(HCV) infection at screening(HCV RNA positive if positive for anti-HCV antibody at screening)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | After induction therapy is completed, Every 6 cycles of maintenance, up to 51 months every 6month
  The percentage of subjects with complete response(CR)
Overall response rate | After induction therapy is completed, Every 6 cycles of maintenance, up to 51 months every 6month

SECONDARY OUTCOMES:
Duration of response | Up to 51 months
Progression free-survival | Up to 51 months
  The time until defined by date of all-cause mortality from the date of investigational procuct administration
Overall survival | the time between the date of treatment start and the date of death due to any cause of disease progression assessed up to 51 months
  It is a measure of the period of survival without disease progression
Time to response | Up to 51 months
Adverse events | From the day 1 of the clinical trial to 28 days after last drug administration
  Investigation of adverse events occurred in subject

CONTACTS AND LOCATIONS:
Locations (1):
- 81, Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul, South Korea